CLINICAL TRIAL: NCT00886938
Title: rTMS To The Dorsolateral Prefrontal Cortex For Patients With Subjective Idiopathic Tinnitus. A Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor, Washington University School of Medicine, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0551
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2012-05-21 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Tinnitus
Keywords: tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Magnetic Stimulation; Pilot Projects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rTMS to DLPF, pilot study (Experimental): rTMS to the dorsolateral prefrontal cortex for patients with tinnitus
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS), pilot study

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS), pilot study — Repetitive transcranial magnetic stimulation, pilot study
  Other Names: Tinnitus; rTMS; Dorsolateral Prefrontal Cortex; DLPF; fcMRI

SUMMARY:
The neurological basis of tinnitus is uncertain when there is no evidence of damage to the peripheral auditory system. However, neuroimaging studies of tinnitus patients show hyperactivity in several cortical regions, especially the auditory cortices and middle temporal regions. A potentially promising treatment modality for tinnitus is repetitive transcranial magnetic stimulation (rTMS). rTMS involves the application of frequent, repeated magnetic stimuli to the skull to induce electrical activity in the underlying cortical areas of the brain. When the magnetic device is placed on the skull, the resultant magnetic field passes through the skull and induces a small secondary current in the cortex. It has been hypothesized that the effect of the frequency used in rTMS differentially influences cortical activity with low-frequency (1Hz) stimulation decreasing and high-frequency stimulation (10-20 Hz) increasing cortical activity.

Currently, reports on treating tinnitus with rTMS have focused on low-frequency stimulation of the left auditory cortex, an area that has been demonstrated to be hyperactive in tinnitus. The benefits of low-frequency auditory cortex stimulation are time limited however. Converging data implicate structures of the brain that are important for mood and attention as playing a role in the maintenance of tinnitus; suggesting an alternative rTMS treatment approach that targets these structures. A growing number of studies demonstrate involvement of the prefrontal cortex in the generation and maintenance of tinnitus. rTMS stimulation in the dorsolateral prefrontal cortex in association with stimulation in the temporoparietal cortex has been shown to increase the durability of the TPC stimulation. The independent effect of rTMS stimulation to the DLPFC is not known. Studies in depression suggest that increasing the intensity and duration of stimulation has beneficial treatment effects. However, the field is new and more work is needed to assess the effectiveness of this treatment, predictors and correlates of response, and safety.

Herein, we propose an open-label pilot study investigating the effectiveness of rTMS stimulation of the dorsolateral prefrontal cortex, an area known to be important for mood and attention, in the treatment of tinnitus

DETAILED DESCRIPTION:
See description above.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18 and 60 years.
* Subjective, idiopathic, troublesome, unilateral or bilateral, non-pulsatile tinnitus of ≥ 6 month's duration..
* Tinnitus handicap score of 38 or greater on the Tinnitus Handicap Inventory.
* Must be able to understand, speak, read, and write English proficiently
* Able to provide informed consent

Exclusion Criteria:

* Patients with tinnitus related to cochlear implantation, retrocochlear lesion, or other known anatomic/structural lesions of the ear and temporal bone. Patients with a history of stapedectomy and insertion of implant may be included if their prosthesis is magnetically safe (MRI compatible up to and including 3T). Patient must be able to provide documentation from surgeon regarding manufacturer information of prosthesis before they will be considered into study.
* Hypersensitive to noises (hyperacusis)
* Patients with cardiac pacemakers; intracardiac lines; implanted medication pumps; implanted electrodes in the brain; other implanted electrical or magnetic medical devices; or other intracranial metal objects or shrapnel, with the exception of dental fillings and MRI compatible stapedectomies or any other contraindication for MRI scan
* Patients with additional significant neurological disorders including increased intracranial pressure, brain mass, epileptic seizures (or family history of epileptic seizures), history of stroke, transient ischemic attack within 2 years, cerebral aneurysm, Huntington's chorea or multiple sclerosis.
* Patients with an acute or unstable medical condition including all patients with any significant heart disease, heart murmur, pneumonia, acute GI bleed, uncontrolled hypertension, or other disorders which would require stabilization prior to initiation of transcranial magnetic stimulation.
* Active alcohol and/or drug dependence or history of alcohol and/or drug dependence within the last year.
* Patients with clinical depression as evidenced by a score of 18 or greater on the Beck Depression Inventory98 or who or, in the opinion of the psychiatric sub-investigator demonstrates active mood symptoms that meet DSM-IV-TR criteria for Major Depressive Disorder
* Patients with psychological illness or trauma which would prohibit participation in the study.
* Female patients of child-bearing potential, unless sterilized or using an appropriate form of birth control acceptable to the research team.
* Currently breastfeeding
* Currently pregnant
* Patients will be excluded if a motor threshold cannot be elicited
* Patients who or are taking over-the-counter or prescribed medication administered for the treatment of any psychiatric or neurologic disorder or any other known CNS active drugs, including herbal, over-the-counter, and homeopathic medications, MAOIs, other antidepressants, antipsychotics, and mood stabilizers.
* Patients whose ability to give informed consent is in question
* Undiagnosed symptomatic hypertension: (for this study defined as systolic blood pressures above 140 mm or diastolic pressure above 90 mm). Subject will be referred to their PCP and not allowed to continue in screening without a note from the PCP stating that they are under his care and have been asymptomatic and with subject's hypertension controlled for at least 3 months.
* Undiagnosed asymptomatic hypertension: (for this study defined as systolic blood pressures above 140 mm or diastolic pressure above 90 mm). Subject will be allowed to continue in the screening process at the discretion of the PI. However, the subject will be referred to his PCP and not allowed to start treatment without a note from his PCP stating that either he was evaluated and his blood

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD,CPI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 06/2009-08/2010 Subjects recruited from Washington University Clinics and from Washington University Volunteers for Health.
Pre-assignment Details: Screening for Motor Threshold with rTMS magnet resulted in screen failure for one subject. Screening for psych history with psychiatrist screen failed one subject. And another subject admitted to falsifying his information, he was withdrawn from the study during screening.
Groups:
- rTMS: rTMS to the dorsolateral prefrontal cortex for patients with tinnitus. Treated at 110% of Motor Threshold
Period: Overall Study
Arm/Group | rTMS
Started | 12
Completed | 10
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | rTMS
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 51 [45 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Average Change (Baseline-End of Treatment) Tinnitus Handicap Inventory (THI)
Description: Patient self-reported Tinnitus Handicap Inventory (THI) The mean change (95% CI) in THI scores (Baseline - End of Treatment). Measures tinnitus severity, or how much tinnitus interrupts their life. The THI scores range from 0-100. 0 being no interruption, 100 being severe interruption in their life from tinnitus.
Time Frame: 0,4 weeks
Population: Total number of participants completing the full four weeks of treatment, according to protocol.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- rTMS: rTMS to the left dorsolateral prefrontal cortex for patients with tinnitus
Arm/Group | rTMS
Number analyzed (Participants) | 10
units on a scale | 10.7 [2.4 to 19]

ADVERSE EVENTS:
Arm/Group | rTMS
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
Open label study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes